CLINICAL TRIAL: NCT04433143
Title: To Evaluate the Efficacy and Safety of Different Intense Pulsed Light Filters Combined With Oral Medication in the Treatment of Moderate to Severe Acne
Brief Title: Evaluate the Efficacy and Safety of Intense Pulsed Light Filters Combined With Oral Medication in the Treatment of Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gang Wang (Other)
Responsible Party: Sponsor-Investigator, Gang Wang, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XijingH-PF-20202021-F-1
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Intense Pulsed Light; Oral Medication
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline; Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral medication (Experimental): just oral minocycline hydrochloride capsules (100mg/ time, once per day),
  Interventions: Drug: Minocycline hydrochloride capsules were taken orally
- Intense Pulsed Light single filter (Experimental): Intense pulsed Acne filter
  Interventions: Drug: Minocycline hydrochloride capsules were taken orally
- Intense Pulsed Light two filters (Experimental): Intense pulsed light Acne filter and another filter (560nm, 590nm or 640nm filter)
  Interventions: Drug: Minocycline hydrochloride capsules were taken orally

INTERVENTIONS:
Drug: Minocycline hydrochloride capsules were taken orally — Lumenis OneTM, OPT tender system produced by American Medical Science Company; Use four of the filters. Acne filter has a wavelength of 400-600/800-1200nm. Three pulses were used for treatment, with a pulse width of 5.0ms, a pulse delay of 30ns, and an energy density of 15j /cm2. The instrument parameters were selected according to the skin lesion characteristics, age and tolerance.
  Other Names: Intense Pulsed Light

SUMMARY:
1. Acne is a chronic inflammatory disease involving the hair follicles and sebaceous glands, characterized by acne, papules, pustules, nodules, and cysts. Acne often occurs in sebum overflow areas such as the face, chest, back and so on. It is a common skin lesion, which not only affects physical health, but also brings psychological disorders and psychosocial problems to patients. At present, the common treatment methods of acne include health education, topical drugs, oral drugs and medical cosmetic treatment.
2. Intense pulsed light has been widely accepted as a non-invasive and non-serious treatment for acne. The M22 strong light and laser system Acne filter has a wavelength of 400-600/800-1200nm.
3. Although there are many treatments for acne, the slow response and easy recurrence of acne are still common problems that trouble doctors and patients. We clinically use drugs combined with intense pulsed light treatment, and the efficacy of the patients is fair, but currently lack of clinical research data support. This study intends to evaluate the effectiveness of different methods in the treatment of moderate and severe acne by evaluating different bands of intense pulsed light combined with drugs, and to observe whether the treatment with oral tetracycline antibiotics combined with intense pulsed light is safe.

DETAILED DESCRIPTION:
The M22 strong light and laser system Acne filter has a wavelength of 400-600/800-1200nm. The light in the 400-600nm band is targeted at the superficial skin inflammation, while 800-1200nm is targeted at the deep sebaceous gland inflammation. The skin can produce oxidation reaction to form singlet oxygen to eliminate propionibacterium acnes after absorption of porphyrin at 400nm. The light of 800-1200nm band can penetrate into the deep layer of sebaceous glands, and the thermal contraction of sebaceous glands can improve the anaerobic environment of bacteria, which is not conducive to the reproduction of bacteria. Meanwhile, when the temperature of sebaceous glands reaches 40 degrees Celsius, bacteria can be killed directly.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40, regardless of gender; The patient agrees to participate in this trial and signs the informed consent Clinical diagnosis of acne (moderate and severe) No bleeding, rupture, infection or other conditions affecting the visual field of laser surgery.

Exclusion Criteria:

* Persons with facial dermatitis and sensitive skin; Relevant treatment within 1 month, including topical drugs, oral drugs, medical cosmetic treatment; Those with a history of exposure to the sun in recent January; Persons with scar constitution; Skin malignant tumor or precancerous lesion; Diabetes, heart disease, epilepsy, connective tissue disease, etc.; Pregnant or breastfeeding; Recent skin infections (such as viruses; Bacteria); Those who are using other methods to treat similar diseases; Others are not suitable for enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-05-06 (Estimated); Study Completion 2021-05-06 (Estimated)

PRIMARY OUTCOMES:
Acne IGA rating scale | change from week0 to week24
  The severity of the facial rash is evaluated according to the number of skin rashes, with a score of 0-5

SECONDARY OUTCOMES:
Pain score | week0，week4，week8
  The pain is rated on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No